CLINICAL TRIAL: NCT06198504
Title: Impact of End-tidal Oxygen Monitoring During Preoxygenation Before Intubation for Acute Hypoxemic Respiratory Failure in ICU Setting: The PFOX Pilot Study.
Brief Title: Impact of End-tidal Oxygen Monitoring During Preoxygenation Before Intubation for Acute Hypoxemic Respiratory Failure in ICU Setting
Acronym: PFOX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC22.0426
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-08

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: Intensive Care Unit (ICU); Intubation; Preoxygenation; End-expiratory tidal oxygen (EtO2)
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Protocol using end-tidal oxygen monitoring during preoxygenation before intubation (Experimental): In 72 consecutive eligible patients tracheal intubation procedure will be performed in accordance with current guidelines except for the duration of the preoxygenation to be individualized by EtO2 monitoring.
  Interventions: Procedure: Protocol using end-tidal oxygen monitoring during preoxygenation before intubation

INTERVENTIONS:
Procedure: Protocol using end-tidal oxygen monitoring during preoxygenation before intubation — According to previous studies a target of EtO2 ≥ 90% is proposed to trigger RSI and intubation. If this target is judged impossible to achieve and/or there is an imperative need to interrupt the pre-oxygenation phase, the operator is free to continue the procedure according to current recommendations.
  Before the start of the inclusions, a training session on the use of the module will be organized with a reminder of the recommendations.
  During the procedure, preoxygenation modalities and duration, achieved EtO2 level, conduction of the induction and intubation, minimum SpO2 and occurrence of complications will be recorded.
  The procedure will stop ten minutes after completion of the orotracheal intubation procedure (defined as inflation of the balloon,clinical and capnography control).

SUMMARY:
The main objective of this pilot study is to determine if our protocole using EtO2 monitoring during preoxygenation before intubation is feasible in a population of critically ill patients in acute hypoxemic respirator failure (AHRF) in Intensive Care Unit (ICU).

We hypothesize that using EtO2 monitoring during preoxygenation before intubation is feasible and safe in a population of critically ill patients in AHRF in ICU setting.

DETAILED DESCRIPTION:
Background : acute hypoxemic respiratory failure (AHRF) is one of the most common causes of intensive care unit (ICU) admission requiring subsequent tracheal intubation for invasive mechanical ventilation. Complications related to tracheal intubation are more frequent in ICU than in operating room with an incidence reaching 20 to 50% in previous studies. Among them, severe hypoxemia and hemodynamic failure can lead to cardiac arrest. End-expiratory tidal oxygen (EtO2) monitoring during preoxygenation is routinely used during anesthesia for elective surgery but has never been evaluated in ICU setting.

Objective : to evaluate the feasibility of a protocol using EtO2 monitoring during preoxygenation before intubation of patients in AHRF in ICU.

Methods : this is an interventional, prospective, bicenter (two French tertiary teaching Hospitals ICUs), feasibility study of a protocol using EtO2 monitoring during preoxygenation before rapid sequence induction (RSI) and intubation of patients in AHRF in ICU. Eligible patients will be older than 18 years, admitted to the ICU, requiring intubation, in AHRF according to the following criteria : a respiratory rate greater than 25 breaths per minute or signs of respiratory distress, and a partial pressure of arterial oxygen (PaO2) to FiO2 ratio equal to or below 200 mmHg (calculation of estimated FiO2 under standard oxygen as follows: FiO2 = 0.21 + oxygen flow rate × 0.03). Main exclusion criteria will be contraindications to Non Invasive Ventilation (NIV) (recent laryngeal, oesophageal, or gastric surgery, and substantial facial fractures), severe haemodynamic failure (Norepinephrine ≥ 0.3 μg/kg/min), cardiac arrest, do not intubate order, pregnancy or breastfeeding and refusal to participate. In 72 consecutive eligible patients tracheal intubation procedure will be performed in accordance with current guidelines except for the duration of the preoxygenation to be individualized by EtO2 monitoring. A targeted EtO2 ≥ 90% will trigger RSI and intubation. During the procedure, preoxygenation modalities and duration, achieved EtO2 level, conduction of the induction and intubation, minimum SpO2 and occurrence of complications will be recorded. A 100- point ponderated score elaborated by an independent expert committee based on literature and updated national guidelines (4,5) will evaluate recommendations adherence. A score ≥ 85 / 100 adjudicates a procedure matching with good practices guidelines. The primary outcome is the percentage tracheal intubation procedures performed in accordance with current good practices guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Admitted in ICU
* In AHRF, defined as : respiratory rate greater than 25 breaths per minute or signs of respiratory distress, and a partial pressure of oxygen (PaO2) to FiO2 ratio equal to or below 200 mmHg (calculation of estimated FiO2 under standard oxygen as follows: FiO2 = 0.21 + oxygen flow rate × 0.03).
* Indication to intubate based on physician judgment
* Written consent obtained from the patient, relative, or emergency consent.

Exclusion Criteria:

* Contraindications to NIV (recent laryngeal, oesophageal, or gastric surgery, and substantial facial fractures)
* Severe haemodynamic failure (Norepinephrine ≥ 0.3 μg/kg/min to maintain MAP ≥ 65 mmHg) or cardiac arrest
* Do not intubate order
* Pregnancy
* breastfeeding
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of tracheal intubation procedures performed in accordance with current good practices guidelines (defined by an independent expert committee score ≥ 85 / 100). | 3 hours

SECONDARY OUTCOMES:
Sequential hierarchical analysis of next criteria | 3 hours
  * Rate of serious complications during procedure defined by following composite criteria : deep hypoxemia (defined by SpO2 < 80%), hemodynamic failure (defined by mean arterial pressure < 65 mmHg despite volume expansion or use of vasopressor), cardiac arrest, death.
  * Rate of moderate complications during procedure defined by composite criteria : hypoxemia (defined by 80% ≤ SpO2 < 90%), difficult intubation (defined as two unsuccessful attempts at laryngoscopy), ventricular or supra-ventricular rhythm trouble, esophageal intubation, aspiration, dental damage.
Duration of preoxygenation | 10 minutes
Maximum EtO2 level achieved | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Florian SIGAUD, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - University Hospital Grenoble, Grenoble
  - University Hospital Lyon, Lyon

REFERENCES:
- [Background] De Jong A, Molinari N, Terzi N, Mongardon N, Arnal JM, Guitton C, Allaouchiche B, Paugam-Burtz C, Constantin JM, Lefrant JY, Leone M, Papazian L, Asehnoune K, Maziers N, Azoulay E, Pradel G, Jung B, Jaber S; AzuRea Network for the Frida-Rea Study Group. Early identification of patients at risk for difficult intubation in the intensive care unit: development and validation of the MACOCHA score in a multicenter cohort study. Am J Respir Crit Care Med. 2013 Apr 15;187(8):832-9. doi: 10.1164/rccm.201210-1851OC. PMID 23348979
- [Background] Nimmagadda U, Salem MR, Crystal GJ. Preoxygenation: Physiologic Basis, Benefits, and Potential Risks. Anesth Analg. 2017 Feb;124(2):507-517. doi: 10.1213/ANE.0000000000001589. PMID 28099321
- [Background] Quintard H, l'Her E, Pottecher J, Adnet F, Constantin JM, De Jong A, Diemunsch P, Fesseau R, Freynet A, Girault C, Guitton C, Hamonic Y, Maury E, Mekontso-Dessap A, Michel F, Nolent P, Perbet S, Prat G, Roquilly A, Tazarourte K, Terzi N, Thille AW, Alves M, Gayat E, Donetti L. Experts' guidelines of intubation and extubation of the ICU patient of French Society of Anaesthesia and Intensive Care Medicine (SFAR) and French-speaking Intensive Care Society (SRLF) : In collaboration with the pediatric Association of French-speaking Anaesthetists and Intensivists (ADARPEF), French-speaking Group of Intensive Care and Paediatric emergencies (GFRUP) and Intensive Care physiotherapy society (SKR). Ann Intensive Care. 2019 Jan 22;9(1):13. doi: 10.1186/s13613-019-0483-1. PMID 30671726
- [Background] Baillard C, Depret F, Levy V, Boubaya M, Beloucif S. Incidence and prediction of inadequate preoxygenation before induction of anaesthesia. Ann Fr Anesth Reanim. 2014 Apr;33(4):e55-8. doi: 10.1016/j.annfar.2013.12.018. Epub 2014 Feb 24. PMID 24582112
- [Background] Samain E, Biard M, Farah E, Holtzer S, Delefosse D, Marty J. [Monitoring expired oxygen fraction in preoxygenation of patients with chronic obstructive pulmonary disease]. Ann Fr Anesth Reanim. 2002 Jan;21(1):14-9. doi: 10.1016/s0750-7658(01)00545-7. French. PMID 11878116
- [Background] Berry CB, Myles PS. Preoxygenation in healthy volunteers: a graph of oxygen "washin" using end-tidal oxygraphy. Br J Anaesth. 1994 Jan;72(1):116-8. doi: 10.1093/bja/72.1.116. PMID 8110535
- [Background] Campbell IT, Beatty PC. Monitoring preoxygenation. Br J Anaesth. 1994 Jan;72(1):3-4. doi: 10.1093/bja/72.1.3. No abstract available. PMID 8110546
- [Background] Frerk C, Mitchell VS, McNarry AF, Mendonca C, Bhagrath R, Patel A, O'Sullivan EP, Woodall NM, Ahmad I; Difficult Airway Society intubation guidelines working group. Difficult Airway Society 2015 guidelines for management of unanticipated difficult intubation in adults. Br J Anaesth. 2015 Dec;115(6):827-48. doi: 10.1093/bja/aev371. Epub 2015 Nov 10. PMID 26556848
- [Background] Tanoubi I, Drolet P, Donati F. Optimizing preoxygenation in adults. Can J Anaesth. 2009 Jun;56(6):449-66. doi: 10.1007/s12630-009-9084-z. Epub 2009 Apr 28. PMID 19399574
- [Background] Caputo ND, Oliver M, West JR, Hackett R, Sakles JC. Use of End Tidal Oxygen Monitoring to Assess Preoxygenation During Rapid Sequence Intubation in the Emergency Department. Ann Emerg Med. 2019 Sep;74(3):410-415. doi: 10.1016/j.annemergmed.2019.01.038. Epub 2019 Mar 14. PMID 30879700
- [Background] Oliver M, Caputo ND, West JR, Hackett R, Sakles JC. Emergency physician use of end-tidal oxygen monitoring for rapidsequence intubation. J Am Coll Emerg Physicians Open. 2020 Sep 28;1(5):706-713. doi: 10.1002/emp2.12260. eCollection 2020 Oct. PMID 33145509
- [Background] Jaber S, Rolle A, Godet T, Terzi N, Riu B, Asfar P, Bourenne J, Ramin S, Lemiale V, Quenot JP, Guitton C, Prudhomme E, Quemeneur C, Blondonnet R, Biais M, Muller L, Ouattara A, Ferrandiere M, Saint-Leger P, Rimmele T, Pottecher J, Chanques G, Belafia F, Chauveton C, Huguet H, Asehnoune K, Futier E, Azoulay E, Molinari N, De Jong A; STYLETO trial group. Effect of the use of an endotracheal tube and stylet versus an endotracheal tube alone on first-attempt intubation success: a multicentre, randomised clinical trial in 999 patients. Intensive Care Med. 2021 Jun;47(6):653-664. doi: 10.1007/s00134-021-06417-y. Epub 2021 May 25. PMID 34032882